CLINICAL TRIAL: NCT01623648
Title: Effect of Whey Protein vs Other Proteins in the Breakfast on Appetite, Overall Postprandial Glycemia and Weight Loss, in Obese Diabetic Individuals
Brief Title: High Protein Breakfast on Appetite, Postprandial Glycemia and Weight Loss in T2D
Acronym: HPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas Caracas (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, MD, MD, Hospital de Clinicas Caracas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCCCBI 017-2007-104
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes
Keywords: whey protein; hunger
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Whey; Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 Whey Breakfast (Experimental): The arm 1 will be assigned to eating Whey protein in the breakfast (660 kcal), lunch (560 cal) and dinner (280 cal), with 42 g protein namely from whey at breakfast
  Interventions: Other: Arm 1 Whey Breakfast
- Arm 2: No Whey Breakfast (Active Comparator): The arm 2 will be assigned to intake other proteins (No Whey) in the breakfast (660 kcal), lunch (560 cal) and dinner (280 cal), with 42 g protein from other sources at breakfast
  Interventions: Other: Arm 2 No Whey Breakfast
- Arm 3: Low Protein Breakfast (Placebo Comparator): The arm 3 will be assigned to intake low protein and high carbohydrate breakfast (660 kcal), lunch (560 cal) and dinner (280 cal), with 22 g protein from other sources at breakfast
  Interventions: Other: Arm 3 Low Protein Breakfast

INTERVENTIONS:
Other: Arm 1 Whey Breakfast — The patients will be assigned to eat 42 g protein namely from Whey protein in the breakfast (660 kcal), lunch (560 kcal) and dinner (280 kcal)
  Other Names: Whey
  Arms: Arm 1 Whey Breakfast
Other: Arm 2 No Whey Breakfast — The patients will be assigned to eat 42 g protein from other sources in the breakfast (660 kcal), lunch (560 kcal) and dinner (280 kcal)
  Other Names: No Whey
  Arms: Arm 2: No Whey Breakfast
Other: Arm 3 Low Protein Breakfast — The patients will be assigned to eat 22 g protein from other sources in the breakfast (660 kcal), lunch (560 kcal) and dinner (280 kcal)
  Other Names: Low Protein
  Arms: Arm 3: Low Protein Breakfast

SUMMARY:
The investigators hypothesis is that eating whey protein in the breakfast versus other proteins will results in higher satiety, reduced overall postprandial glycemia and more weight loss in obese diabetic individuals

DETAILED DESCRIPTION:
Recently we have shown that compared to low carbohydrate diet, an isocaloric diet with addition of high calorie and protein breakfast promoted sustained weight loss and prevented weight regain by reducing diet-induced compensatory changes in hunger, cravings and ghrelin suppression.

However the effect of isocaloric and isoproteic breakfast with different source of proteins, (whey vs other proteins or vs low protein in breakfast) on weight loss, appetite and on glycemic fluctuations after breakfast lunch and dinner was not explored in obese diabetic individuals.

To search whether compared to proteins like tuna, eggs and soy, the intake of whey protein in the breakfast will lead to reduced hunger and overall postprandial glycemia and will enhance weight loss in obese diabetic individuals

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥30 and ≤70 years of age
2. BMI: 26 to 34 kg/m2)
3. Diabetes criteria
4. HbA1C: 7-9 % or
5. Habitually eat breakfast
6. Only naïve or treated with metformin.
7. Those with anti-hypertensive and lipid-lowering medication will be included.
8. . Not dieting and no change in body weight >10 lb = 4.5 kg within the last 6 months

10.Those who provide signed informed consent 11.Stable physical activity pattern during the three months immediately preceding study initiation.

12. Normal liver, kidney and thyroid function. 13. Negative urinary microalbumin test (urMA) and estimated glomerular filtration rate (GFR) > 60 mL/min/1.73 m2.

Exclusion Criteria:

1. Type 1 Diabetes
2. Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, malignant disease
3. Anemia (Hg > 10 g/dL)
4. Serum creatinine level < 1.5 mg/dl
5. Pulmonary disease, psychiatric, immunological, neoplastic diseases or severe diabetic complications, such as cardiovascular disease, cerebrovascular disease, proliferative diabetic retinopathy, gastroparesis or underwent bariatric surgery.
6. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase and/or aspartate
7. Infectious disease
8. Malignancy
9. Pregnant women or lactating
10. Known hypersensitivity to milk components

10. Participating in dietary program or using of weight-loss medications 11. Documented or suspected history (within one year) of illicit drug abuse or alcoholism.

12. Use of psychotropic, anorectic or steroid medication during the month immediately prior to study onset

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | 12 weeks
  Postprandial plasma glucose after breakfast, lunch and dinner

SECONDARY OUTCOMES:
Plasma Insulin | 12 weeks
  Postprandial plasma insulin after breakfast lunch and dinner
Hunger | 12 weeks
  Postprandial Hunger after breakfast lunch and dinner, assessed with visual analog scale.
Satiety | 12 weeks
  Postprandial Satiety after breakfast lunch and dinner, assessed with visual analog scale.
Change in body weight | 12 weeks
  Body weight will be assessed every every two weeks until week 12

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Hospital de Clinicas Caracas
Locations (2):
- Daniela Jakubowicz, Holon, N/A = Not Applicable, Israel
- Daniela Jakubowicz, Caracas, San Bernardino, Venezuela